CLINICAL TRIAL: NCT05274711
Title: The Effect of Whole Body Vibration on Neck Disability and Proprioception in Patients With Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ali Saaid Mahmoed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003408
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Intervention Model Description: This trail has 2 groups one control and one experimental
Who Masked: Investigator, Outcomes Assessor
Masking Description: Opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): will receive conventional physical therapy prograM
  Interventions: Other: Conventional physical treatment
- Experimental treatment (Experimental): will receive conventional physical therapy program and whole body vibration training
  Interventions: Other: Whole body vibration training; Other: Conventional physical treatment

INTERVENTIONS:
Other: Whole body vibration training — The participants will be instructed to stand on the vibration platform bare footed and distribute their weight evenly on both feet (fig 3). Next, they will be asked to do a head and neck retraction while looking forward with their knees at 30 degrees of flexion. In order to prevent fatigue in the subject's cervical area due to holding their head and neck in retraction, they will be asked to hold this position for 15 seconds then rest for 5 seconds. Since each set will last 60 second this allowed the subjects to do 3 retractions in each set. In total each subject will perform 15 retractions during the training. The subjects will experience a vertical vibration at a frequency and amplitude of 30 Hz and 4 mm during the sets (Salami et al., 2018).
  Arms: Experimental treatment
Other: Conventional physical treatment — Posturalcorrectionexercisesintheformofstretchingandstrengthening exercise. Manual stretching exercises as passive stretch to (upper trapezius, levator scapulae, sub occipitalis, scalene, sternocleidomastoid, and pectoralis major muscles), 30 seconds of 3-5 repetitions for each muscle, followed by 30 seconds of rest, as well as isotonic exercises (to strength deep neck flexors and scapular retractor muscles) 3 sets of 12 repetitions each with a 6 second hold in between, with a 1-2-minute rest between sets (Kisner. and Colby 2012).

SUMMARY:
To investigate if the Whole-body vibration affect cervical function cervical, proprioception, pain intensity level and ROM and in subjects with forward head posture?

DETAILED DESCRIPTION:
Forward head posture (FHP) is one of the most common types of postural abnormality, and it is generally described as an anterior position of the head in relation to the vertical line of the body's center of gravity. Many researchers have reported that several factors, including headache, neck pain, and musculoskeletal disorders such as temporomandibular disorders or rounded shoulders, are related to FHP In forward head posture (FHP) lower cervical vertebrae are bent and upper cervical vertebrae are extended, and the weight of the head supported by the neck is increased. The bending moment of the head applies pressure on muscles and joints around the cervical vertebrae, in addition to active myofascial trigger points of the suboccipital muscle which may induce tension type headaches, neck pain and cervical headaches, while reducing the mobility of the neck Furthermore, FHP was associated with shortening of the upper trapezius, the posterior cervical extensor muscles, the sternocleidomastoid muscle and the levator scapulae muscle Recently studies have reported impaired proprioception to be one of the results of prolonged FHP. The cervical spine proprioceptive system is responsible for head orientation in space and in relation to the trunk and it is known for its role in maintaining head and neck stability It was concluded that the craniovertebral angle (CVA) is negatively correlated with the disability of patients with neck pain. So, patients with small CVA have a greater forward head posture, and the greater the forward head posture, the greater the disability.

Neck pain is a common complaint in the population. It has an episodic occurrence with variable recovery between episodes, and it is considered the most persistent musculoskeletal pain syndrome. Regarding physical work factors, neck pain was significantly associated with holding the neck in a forward bent posture for a prolonged time and making repetitive movements Despite claims that FHP may be related to neck pain, existing evidence seems controversial, since some previous studies have reported no significant associations between neck pain and FHP whereas other studies have reported an association between FHP and neck pain. It was showed that adults with neck pain have significantly more FHP than asymptomatic adults. Greater FHP has been associated with greater deficits in cervical range of motion, particularly neck rotation and flexion. Also, FHP seems to have a negative impact on static balance control in asymptomatic adults.

Corrective exercise is one of the interventional methods that had been suggested for treatment of FHP, including stretching, strengthening, and movement control exercises. Moreover, there may be advantages in exercising adjacent body segments to the cervical spine, such as the thoracic spine, to enhance the effectiveness of exercise training on FHP. Several studies have shown that corrective exercise regimes can improve FHP and potentially related symptoms. For example, exercise training protocols have resulted in improvement of CVA, head tilt, cranial or cervical range of motion neck disability and pain

Whole-body vibration exercise (WBV) may enhance muscle strength adaptations associated with traditional neuromuscular training or rehabilitation. The potentially beneficial effects of WBV are caused by the transmission of mechanical, sinusoidal vibrations throughout the body via the feet WBV is a neuromuscular training method that has recently been developed. In WBV training, the subject stands on a platform that generates vertical sinusoidal vibration at a frequency between 35 and 40 Hz. These mechanical stimuli are transmitted to the body where they stimulate in turn sensory receptors, most likely muscle spindles. This leads to the activation of the alpha-motoneurons and initiates muscle contractions comparable to the earlier described "tonic vibration reflex" Whole-body vibration (WBV) has become increasingly popular with reports of improved strength, power, movement velocity as well as balance and flexibility (Pollock et al., 2010). WBV exercises are performed while standing on a motor driven oscillating platform device. The mechanical vibration stimulus applied to the muscles and tendons during WBV exercise is characterized by a cyclic transition between eccentric and concentric muscle contractions and leads to a neuromuscular response

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent physical therapy students of both gender between 18-23 years old
2. BMI between 18.5-25 kg/m²
3. Symptomatic forward head posture with CVA 49° or less.

Exclusion Criteria:

1. Cervical disc
2. Myelopathy or cervical radiculopathy
3. Cervical spine surgery in the past
4. Having received physical therapy in the three months prior to the study

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The change in Neck disability | immediately after the treatment
  Neck disability will be measured by English neck disability index (NDI) questionnaire is composed of a total of 10 questions. Each question has 6 answer options which pertain to a level of severity (0-5) With total score of 50 , when NDI is high the neck function is the worst
The change in Neck proprioception | immediately after the treatment
  Neck proprioception will be measured by clinometer application

SECONDARY OUTCOMES:
Neck pain | Before and immediately after the treatment
  Neck pain will be measured be visual analogue scale (VAS). When responding to a VAS item, patients make marks along the 100 mm line at the point they feel represents their current pain state. With 100 mm means high level of pain and 0 means no pain
Cervical ROM | Before and immediately after the treatment
  Cervical ROM will be measured by clinometer application

CONTACTS AND LOCATIONS:
Locations (1):
- Aya Ali saaid mahmoed, Cairo, Egypt